CLINICAL TRIAL: NCT06596850
Title: Efficacy of Wheelchair Skills Training to Improve Mobility for People with ARSACS and DM1
Brief Title: Wheelchair Skills Training for People with ARSACS and DM1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-3100
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Wheelchair Mobility; Manual Wheelchair Skills Training; ARSACS; Myotonic Dystrophy Type 1
MeSH Terms: conditions — Spastic ataxia Charlevoix-Saguenay type; Myotonic Dystrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wheelchair Skills Training Program (WSTP) (Experimental): Standardized wheelchair skills training program.
  Interventions: Behavioral: Wheelchair Skills Training Program
- Control (No Intervention): Wait-list control group where participants will receive usual care from their clinician.

INTERVENTIONS:
Behavioral: Wheelchair Skills Training Program — Participants will receive 5, 45-minute weekly WC skills training sessions that will take place in the community, in and around the participants home. Each session will be customized to the participant's' goals and based on the learner's impairments (i.e., weakness, spasticity, movement disorders [e.g. ataxia, tremor], contractures, cognition). The WSTP sessions will begin with a 5-minute review of goals/progress, followed by a 10-minute warm-up (wheeling activities, random practice of previously leaned skills); 20 minutes of attempting new skills (training on each skill will be carried to next session until the skills are learned or until the trainer and participant mutually agree that training should be abandoned; the trainer will periodically ask the participant to practice newly learned skills to incorporate variability of practice); 10 minute cool-down, during which the participant will practice skills in a self-controlled environment.
  Arms: Wheelchair Skills Training Program (WSTP)

SUMMARY:
Wheelchairs (WC) are often provided to people with ARSACS and MD1 when they are not able to walk anymore. However, giving someone a MWC alone does not guarantee they will use it safely or properly. Many people who use WC need help from others to get around and they can not always do the things they like to do. This can lead to isolation, stress, and reduced quality of life. In addition, poor use of a MWC could lead to accidents and injuries. Our team recently showed that people with ARSACS have lower MWC skills than other adults who use MWC, and that teaching MWC skills to people with ARSACS seems to work. Now we are ready to test the program with more people with ARSACS and MD1 to see how it can improve MWC mobility and confidence. We also want to hear about people's expectations and experiences with MWC training. People who take part in research will answer questions before and after WC training, and we will follow up with them 3 months later to ask again about their WC use.

This projects directly adresses the mobility needs of people with ARSACS and MD1 who use MWC. Our results may improve how therapists provide training for MWC use, which may improve mobility, participation, and quality of life for people with ARSACS and MD1. Learning just one MWC skill could be life-changing. It could mean the difference between leaving the house or not, which could impact the ability to shop for groceries, see friends, or to have a job.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age, have a diagnosis of ARSACS or DM1, and use a manual WC for mobility (≥3 times/week for ≥8 hours/week).

Exclusion Criteria:

* anticipate a health condition or procedure that contraindicates training (e.g., surgery); or concurrently or planning to receive WC training during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Wheelchair Skills Test Questionnaire (WST-Q) | Baseline (T1); immediately post intervention up to 5 weeks after baseline (T2); 3-months follow-up (T3)
  Subjective report of participants' perceived manual wheelchair skills (performance and frequency). The WST-Q comprises 30 discrete manual WC skills. Skills are scored on a scale ranging from 0 (cannot execute skill) to 3 (can execute skill with expertise); a total percentage score (0-100%) is calculated with higher scores representing greater wheelchair skills. The WST-Q can be completed in ~15 minutes, has strong psychometric properties in English and French, and has been used extensively in clinical trials. The WST-Q has been validated by the study team for ARSACS.

SECONDARY OUTCOMES:
Wheelchair Skills Test (WST) | Baseline (T1); immediately post intervention up to 5 weeks after baseline (T2); 3-months follow-up (T3)
  Objective rating of participants' perceived manual wheelchair skills (capacity). The WST comprises 30 discrete manual WC skills. Skills are scored on a scale ranging from 0 (cannot execute skill) to 3 (can execute skill with expertise); a total percentage score (0-100%) is calculated with higher scores representing greater wheelchair skills. The WST-Q can be completed in ~30 minutes, has strong psychometric properties in English and French, and has been used extensively in clinical trials. The WST-Q has been validated by the study team for ARSACS.
Wheelchair Use Confidence Scale (WheelCon) | Baseline (T1); immediately post intervention up to 5 weeks after baseline (T2); 3-months follow-up (T3)
  WC use confidence (i.e., belief in ability to accomplish specific tasks while using a manual WC) will be assessed using the Wheelchair Use Confidence Scale for Manual Wheelchair Users Short Form (WheelCon-M). The WheelCon-M comprises 21 statements related to confidence using a MWC in activities and environments, each rated on a scale from 0 ("not confident") to 10 ("completely confident"), producing a total mean score between 0 and10. Higher scores represent higher confidence. The WheelCon-M was validated for ARSACS.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Interdisciplinary Research in Rehabilitation and Social Integration, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niyomwungere E, Routhier F, Gagnon C, Kirby RL, Rodrigue X, Lessard I, Lettre J, Best KL. Efficacy of Manual Wheelchair Skills Training for Improving Skills and Confidence in People With Hereditary Degenerative Disorders: Protocol for a Sequential Multimethods Study. JMIR Res Protoc. 2025 Jul 31;14:e66974. doi: 10.2196/66974. PMID 40742628